CLINICAL TRIAL: NCT05381974
Title: The Effects of Psilocybin on Self-Focus and Self-Related Processing in Treatment Resistant MDD
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to difficulty recruiting patients who met inclusion/exclusion criteria. No participants received the intervention.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: COMPASS Pathways (Industry)
Responsible Party: Principal Investigator, Sharmin Ghaznavi, Psychiatrist, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2021P000863
Record Dates: First submitted 2022-05-10; First posted 2022-05-19 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Treatment-Resistant Major Depressive Disorder
Keywords: Psilocybin; Neuroimaging; Rumination; Treatment-Resistant Depression
MeSH Terms: conditions — Rumination Syndrome; Depressive Disorder, Treatment-Resistant | interventions — Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Psilocybin (Experimental): 25mg of Psilocybin
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — Open-Label

SUMMARY:
This open-label fMRI study will assess the effects of a single dose of psilocybin on rumination and the neural correlates of rumination in individuals with treatment-resistant major depressive disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Must be able to sign the informed consent form (ICF).
2. Be 18-55 years of age at screening.
3. At least moderate MDD based on clinical assessment and a structured clinical interview, the Mini International Neuropsychiatric Interview Version 7.02 (MINI).
4. Hamilton Depression Rating Scale - 17 item (HAM-D-17) score ≥ 18 at Screening and at Baseline.
5. Failure to respond to an adequate dose and duration of 2, 3, or 4 pharmacological treatments for the current episode as determined through the Massachusetts General Hospital Antidepressant Treatment History Response Questionnaire (MGH-ATRQ) and using the supplementary advice on additional antidepressants not included in MGH-ATRQ. Augmentation with an add-on treatment counts as a second treatment, provided it is approved for the adjunctive treatment of MDD.
6. McLean Screening Instrument for Borderline Personality Disorder (MSI-BPD) < 7 at Screening.
7. Have successfully discontinued all antidepressant medications at least 2 weeks prior to Baseline Scan. (Please note: once enrolled in the study, participants will have to successfully undergo a taper off of all psychotropic medications under the supervision of a study psychiatrist and in coordination with their treatment team).
8. A score > 40 on the Wechsler Test of Adult Reading.
9. Be right-handed as determined by the Edinburg Handedness Inventory.
10. Ability to complete all protocol required assessment tools without any assistance or alteration to the copyrighted assessments, and to comply with all study visits.
11. Have ongoing established mental health care.

Exclusion Criteria:

1. Current, past history, or family history, of schizophrenia, psychotic disorder (unless substance induced or due to a medical condition), bipolar disorder, delusional disorder, paranoid personality disorder, schizoaffective disorder, borderline personality disorder, or any serious psychiatric comorbidity as assessed by medical history and a structured clinical interview (version 7.0.2 MINI).
2. Positive MR screen (e.g., metal implant, claustrophobia, etc).
3. Prior electroconvulsive therapy and/or ketamine for current episode.
4. Current cognitive behavioral therapy (CBT) that will not remain stable for the duration of the study. CBT cannot be initiated within 21 days of Baseline.
5. Current (within the last year) alcohol or substance abuse as informed by DSM-5 at Screening.
6. Significant suicide risk as defined by (1) suicidal ideation as endorsed on items 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) within the past year, at Screening or at Baseline, or; (2) suicidal behaviors within the past year, or; (3) clinical assessment of significant suicidal risk during clinical interview.
7. Significant homicide risk as defined by clinical interview.
8. Depression secondary to other severe medical conditions.
9. Currently taking benzodiazepines daily.
10. Other personal circumstances and behavior judged to be incompatible with establishment of rapport or safe exposure to psilocybin, as well as exposure to psilocybin or other psychedelics within one year of screening.
11. Women who are pregnant, nursing, or planning a pregnancy. Participants who are sexually active must agree to use a highly effective contraceptive method throughout their participation in the study. Women of childbearing potential must have a negative urine pregnancy test at Screening and Day Before Psilocybin.
12. Cardiovascular conditions: recent stroke (< 1 year from signing of consent), recent myocardial infarction (< 1 year from signing of ICF), hypertension (blood pressure > 140/90 mmHg) or QTc > 450 msec) or clinically significant arrhythmia within 1 year of signing the ICF, current anticoagulant therapy, aneurysmal disease.
13. Uncontrolled insulin dependent diabetes.
14. Seizure disorder.
15. Positive urine drug screen for illicit drugs or drugs of abuse (to include but not limited to opiates, PCP, cocaine, amphetamines, methamphetamines, benzodiazepines, barbiturates, and cannabis) at Screening and Day Before Psilocybin. Any positive urine drug test will be reviewed with participants to determine the pattern of use and eligibility will be determined at the investigator's discretion.
16. Lifetime history of surgical procedures involving the brain or meninges, encephalitis, meningitis, degenerative central nervous system (CNS) disorder (e.g., Alzheimer's or Parkinson's Disease), epilepsy, mental retardation, or any other disease/procedure/accident/intervention which, according to the screening clinician, is deemed associated with significant injury to or malfunction of the CNS, or history of significant head trauma within the past 2 years.
17. Any current or past history of any physical condition which in the investigator's opinion might put the subject at risk or interfere with study results interpretation.
18. Current enrollment in any investigational drug or device study or participation in such within 6 months of Screening.
19. Current enrollment in an interventional study for depression or participation in such within 6 months of Screening Visit.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Change in Massachusetts General Hospital Rumination Questionnaire (MGH-RQ) | Baseline, and 3 weeks, 6 weeks, 9 weeks, and 12 weeks after psilocybin administration.
  A transdiagnostic state measure of rumination over the previous two weeks consisting of 9 items on a 5 point Likert scale from 0 (Never/Rarely) to 4 (All The Time).
Change in Resting-State Functional Connectivity | Baseline, day of psilocybin administration, and 3 weeks, and 12 weeks after psilocybin administration.
  Changes in resting-state activity during functional magnetic resonance imaging(fMRI) scans.
Change in Self-Attribution Task performance | Baseline, day of psilocybin administration, and 3 weeks, and 12 weeks after psilocybin administration.
  Participants are shown words one at a time and asked to answer if each of the words apply to 'Self' or 'Other'
Change in Task-Based Activity during Self-Attribution Task | Baseline, day of psilocybin administration, and 3 weeks, and 12 weeks after psilocybin administration.
  Changes in task-based activity during functional magnetic resonance imaging(fMRI) scans.

SECONDARY OUTCOMES:
Change in Montgomery-Asberg Depression Rating Scale(MADRS) | Baseline, the day before psilocybin administration and at 1 day, 1 week, 2 weeks, 3 weeks, 6 weeks, 9 weeks and 12 weeks after psilocybin administration.
  The MADRS is a clinician-rated scale measuring depression severity, consisting of 10 items, each scored from 0 (normal) to 6 (severe), for a total possible score of 60; higher scores denote greater severity.
Change in Quick Inventory of Depressive Symptomatology - 16 item (QIDSR-SR-16) | Baseline, the day before psilocybin administration and at 1 day, 1 week, 2 weeks, 3 weeks, 6 weeks, 9 weeks and 12 weeks after psilocybin administration.
  The 16-item QIDS-SR-16 a self-rated scale designed to assess the severity of depressive symptoms in the nine diagnostic symptom domains of a major depressive episodes, exclusive of atypical or melancholic symptoms. The QIDS-SR-16 is sensitive to change with various treatments, demonstrating its utility in research settings. The total score ranges from 0 to 27 with 0 representing no depression and 27 representing severe depression.
Change in Positive and Negative Affect Schedule (PANAS) | Baseline, the day of psilocybin administration and at 3 weeks and 12 weeks after psilocybin administration.
  The PANAS measures the acute emotional drug effects and comprises 2 mood scales that measure positive and negative affect. Participants respond to 20 items using a 5-point scale that ranges from "slightly or not at all (1)" to "extremely (5)". A total higher score on the positive affect questions indicates more of a positive affect while a lower score on the negative affect questions indicates less of a negative affect.
Change in Hamilton Depression Rating Scale - 17 item (HAM-D-17) | Baseline and 3 weeks and 12 weeks after psilocybin administration.
  The HAM-D-17 is a 17 item scale used to assess the degree of symptom severity in depressed patients.
Change in Ruminative Response Scale (RRS) | Baseline and 12 weeks after psilocybin administration.
  A self-report measure of describing one's responses to depressed mood, consists of 22 items and three factors (Depression, Brooding, and Reflection). Each item is rated on a 4-point Likert scale ranging from 1 (never) to 4 (always). The total score ranges from 22 to 88, with higher scores indicating higher tendency to ruminate, i.e. higher trait rumination.
Change in Rumination Reflection Questionnaire (RRQ) | Baseline and 12 weeks after psilocybin administration.
  The RRQ measures the extent to which a person tends to ruminate or engage in self-reflection. It consists of 24 items measured on a 5 point Likert scale from 1 (Strongly Disagree) to 5 (Strongly Agree),12 items which assess the tendency to ruminate, and 12 items which assess the tendency to engage in self reflection.
Change in Penn State Worry Questionnaire (PSWQ) | Baseline and 12 weeks after psilocybin administration.
  The PSWQ is a 16-item questionnaire that aims to measure the trait of worry, using Likert rating from 1 (not at all typical of me) to 5 (very typical of me). The PSWQ attempts to measure the excessiveness, generality, and uncontrollable dimensions of worry.
Change in NEO-Five-Factor Inventory (NEO-FFI) | Baseline and 12 weeks after psilocybin administration.
  The NEO-FFI is a 60-item psychological personality inventory that assesses based on the five- factor model: Openness to Experience, Conscientiousness, Extraversion, Agreeableness, and Neuroticism. Participants are asked to select the response that best represents their opinion on a 5-point scale: 0-Strongly Agree, 1-Agree, 2-Neutral, 3-Disagree, 4-Strongly Disagree.
Change in Behavior Rating Inventory of Executive Function - Adult Version (BRIEF) | Baseline and 12 weeks after psilocybin administration.
  The BRIEF is a 75-item scale designed to assess executive function and self-regulation. Participants choose how often certain behaviors were problematic over the past month N-never, S-sometimes, O-often.
Change in Cognitive Flexibility Inventory (CFI) | Baseline and 12 weeks after psilocybin administration.
  The CFI is a brief self-report measure of the type of cognitive flexibility necessary for individuals to successfully challenge and replace maladaptive thoughts with more balanced and adaptive thinking. The measure consists of 20 items and participants indicate the extent to which they agree or disagree with the statements in the items, on a scale from 1-Strongly Disagree to 7-Strongly Agree.
Change in Emotional Faces Flanker Task | Baseline, day of psilocybin administration, and 3 weeks and 12 weeks after psilocybin administration.
  This task examines executive functioning as it assesses the ability to ignore/inhibit irrelevant flanking information in order to respond to the central task.
Change in Depression Implicit Attitudes Task (IAT) | Baseline, day of psilocybin administration, and 3 weeks and 12 weeks after psilocybin administration.
  The IAT provides a measure of the strength of association between four categories by pairing two concept categories (e.g., Me/Not-Me) with two attribution categories (e.g., Happy/Sad).

OTHER OUTCOMES:
Change in Social Adjustment Scale-Self-Report - Short Version (SAS-SR: Short) | Baseline and 2 weeks, 3 weeks, and 12 weeks after psilocybin administration.
  The SAS-SR: Short is a 24-item self-report scale rated on a 5-point scale designed to measure social adjustment over the last two weeks.
Change in UCLA Loneliness Scale | Baseline and 2 weeks, 3 weeks, and 12 weeks after psilocybin administration.
  The UCLA Loneliness Scale is a 20-item self-report measure of loneliness. Participants are asked to indicate how often they feel the way described, on a scale from 1-Never to 4-Always.
Change in Brief Fear of Negative Evaluation Scale - Second Version (BFNE-II) | Baseline and 2 weeks, 3 weeks, and 12 weeks after psilocybin administration.
  The BNFE-II is a 12-item self-report measure of social anxiety. Participants are asked to rate how characteristic each statement is of them on a scale from 1-Not at all characteristic of me to 5-Extremely characteristic of me.
Change in Social Provisions Scale (SPS) | Baseline and 2 weeks, 3 weeks, and 12 weeks after psilocybin administration.
  The SPS is a 24-item self-report measure of perceived social support. Participants are asked to rate the extent to which they agree that each statement describes their current relationships with other people on a scale from 1-Strongly Disagree to 4-Strongly Agree.
Change in Self-Consciousness Scale (SCS) | Baseline and 2 weeks, 3 weeks, and 12 weeks after psilocybin administration.
  The SCS is a 22-item self-report measure of private and public self-consciousness as well as social anxiety. Participants are asked to indicate the extent to which each statement is like them on a scale from 0-Not at all like me to 3-A lot like me.
Change in Personal Space Task | Baseline and 3 weeks and 12 weeks after psilocybin administration.
  The Stop Distance Procedure (SDP) will be completed in a virtual reality environment to measure personal space size and permeability.

CONTACTS AND LOCATIONS:
Overall Officials: Sharmin Ghaznavi, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Athinoula A. Martinos Center for Biomedical Imaging, Charlestown, Massachusetts, United States